CLINICAL TRIAL: NCT02885558
Title: Role of T-type Calcium Channels in Vascular Function
Brief Title: Role of Calcium Channels in Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Stefan Mortensen, Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 47880
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Endothelium, Vascular
Keywords: Receptors, Calcium Channel Blocker
MeSH Terms: interventions — efonidipine; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L + T-type (Experimental): 8 weeks treatment with efonidipine (1 week 1x20mg, 7 weeks 2x20mg)
  Interventions: Drug: Efonidipine
- L-Type (Active Comparator): 8 weeks treatment with nifedipine (1 week 1x20mg, 7 weeks 2x20mg)
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Efonidipine — 8 weeks treatment with either efonidipine
  Other Names: Landel (efonidipine)
  Arms: L + T-type
Drug: Nifedipine — 8 weeks treatment with either nifedipine
  Other Names: Adalat (nifedipine)
  Arms: L-Type

SUMMARY:
The purpose of this study is to examine the role of T-type calcium channels in endothelial dysfunction observed with ageing.

ELIGIBILITY:
Inclusion Criteria:

* age 20 - 30 and 60-70
* BMI < 30

Exclusion Criteria:

* Hypertension (>150/90 mmHg)
* Smoking
* Physical activity >2 hours/week
* Known chronic diseases
* Pregnancy or birth within 3 month
* Alcohol misuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Vascular function | 8 weeks
  Hemodynamic response to femoral arterially infused vasoactive substances

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Centre for Phsical Activity Research, Copenhagen
  - Cardiovascular and Renal Research, Odense